CLINICAL TRIAL: NCT02197442
Title: An Open Label, Balanced, Randomized, Two-treatment, Four-period, Two-sequence, Single Oral Dose, Crossover, Fully Replicate Bioequivalence Study of Two Formulations of Valsartan 320 mg Tablet in Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Valsartan 320mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 044-14
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Valsartan Tablets USP 320 mg DIVIS
  Interventions: Drug: Valsartan
- Reference (Active Comparator): Diovan® (Valsartan) 320 Tablets
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan
  Other Names: 320mg tablets

SUMMARY:
The study was an open label, balanced, randomized, two-treatment, four-period, two sequence, single oral dose, crossover, fully replicate bioequivalence study of two formulations of Valsartan 320 mg under fasting conditions.

DETAILED DESCRIPTION:
Tablet in healthy, adult human subjects under fasting condition, with a screening period of 28 days prior to dose administration in Period-I. In each study period, twenty-four (24) blood samples, including two (02) predose blood samples, each of 02 mL were collected from each subject except for the discontinued / withdrawn subjects to analyze the pharmacokinetic profile of the test as well as the reference product.

The pharmacokinetic parameters were calculated from the drug concentration vs. time profile by non-compartmental model using WinNonlin Professional Software-Version 5.3 (Pharsight Corporation, USA) for Valsartan. Statistical comparison of the pharmacokinetic parameters of the two formulations was carried out using PROC MIXED of SAS® Version 9.3 (SAS Institute Inc., USA) to assess the bioequivalence of both the formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, human volunteers between 18 to 45 years of age (both inclusive) living in and around Ahmedabad city or western part of India.
2. Having a Body Mass Index (BMI) between 18.5-24.9 (both inclusive), calculated as weight in kg/height in meter2.
3. Not having any significant disease in medical history or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12- lead ECG and X-ray chest (P/A view) recordings.
4. Able to understand and comply with the study procedures, in the opinion of the investigator.
5. Able to give voluntary written informed consent for participation in the trial.
6. In case of female subjects:

   * Surgically sterilized at least 6 months prior to study participation; Or
   * If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And

• Pregnancy test must be negative.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to valsartan or any of the formulation excipients or any related drug.
2. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
3. Sitting blood pressure less than 110 /70 mm Hg and pulse rate less than 60 or more than 100 beats per minute at the time of screening.
4. Presence of orthostatic hypotension.
5. If the QTc interval were to be more than 450 ms on ECG measurement at the time of screening.
6. Inability to remain in an upright position at the time of dosing.
7. Ingestion of a medicine (including herbal remedies) at any time within 14 days before dosing in period-I. In any such case subject selection were at the discretion of the Principal Investigator.
8. Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
9. A recent history of harmful use of alcohol (less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to receiving study medicine.
10. Smokers, who smoke 10 or more than 10 cigarettes/day or inability to abstain from smoking during the study.
11. The presence of clinically significant abnormal laboratory values during screening.
12. Use of any recreational drugs or history of drug addiction or testing positive in pre study drug scans.
13. History or presence of psychiatric disorders.
14. A history of difficulty in donating blood.
15. Donation of blood (1 unit or 350 mL) or receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study.

    Note: In case the blood loss is ≤ 200 mL; subject may be dosed 60 days after blood donation or last sample of the previous study.
16. A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.
17. A positive test result for HIV antibody.
18. An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medicine in period-I. In any such case subject selection were at the discretion of the Principal Investigator.
19. Consumption of grapefruit or grapefruit products within 48 hours prior to dosing.
20. Nursing mothers (females).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Valsartan | 0-36 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Lambda Therapeutic Research Ltd.,, Ahmedabad, Gujarat, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm